CLINICAL TRIAL: NCT03226574
Title: A Multicenter, Open-Label, Phase 1b Study to Assess the Safety and Define the Maximally Tolerated Dose of Epidural Resiniferatoxin Injection for the Treatment of Intractable Pain Associated With Cancer
Brief Title: Study to Evaluate Safety and MTD of Epidural Resiniferatoxin Injection for Treatment of Intractable Cancer Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTX-001
Record Dates: First submitted 2017-07-06; First posted 2017-07-24 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Intractable Cancer Pain
Keywords: Resiniferatoxin; RTX; Cancer pain
MeSH Terms: conditions — Cancer Pain | interventions — resiniferatoxin

STUDY DESIGN:
Intervention Model Description: The design uses a traditional "3+3" rule-based design that does not stipulate any prior assumption of the dose-toxicity curve. Dose escalation is permitted between successive cohorts based upon a specified algorithm, using discrete dosage steps.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RTX epidural injection (Experimental): Epidural injection of 1.5mL/min RTX under the guidance of epidurogram.
  Interventions: Drug: Resiniferatoxin

INTERVENTIONS:
Drug: Resiniferatoxin — single dose (0.4, 1, 2, 4, 8,15, 25 or 35 mcg), epidural injection
  Other Names: RTX

SUMMARY:
The study is a multicenter, open-label Phase 1b single dose escalation safety study for adult subjects with intractable pain associated with cancer in any area below the mid-thoracic level who meet all other eligibility criteria.

DETAILED DESCRIPTION:
All subjects who received RTX will be included in the analyses and summaries of safety, efficacy, PD, and PK assessments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced cancer or metastasis, which has not responded to standard therapy, producing intractable chronic pain in any area below the mid-thoracic level.
* Male or female subjects must be at least 18 years of age.
* Must have a worst pain score ≥6 on the NPRS at Screening visit.
* Subjects not seeking or receiving potentially curative therapies for cancer. Palliative therapy is acceptable if the therapy started and is stable prior to IP administration.
* Sexually active female subjects of childbearing potential and male subjects capable of fathering a child must be willing to use an effective method of contraception to avoid pregnancies.
* Must be willing and capable of understanding and cooperating with the requirements of the study.
* Must be able to understand and complete study-related forms and adequately communicate with the investigator and/or site staff.
* Must have provided written informed consent prior to participating in any study-related activity.
* Subjects able to complete the study duration.

Exclusion Criteria:

* Subjects with leptomeningeal metastases in lumbar area.
* Undergoing or have plans to undergo changes to current cancer treatment during the study through the Day15 assessment.
* Had prior lumbar spine surgical procedures that could impair the ability to perform the injection.
* Evidence of brain pathology or increase intracranial pressure.
* Presence of an IT shunt.
* Has evidence or a coagulopathy or hemostasis problem.
* Subjects with a total neutrophil count <1500 cells/mm3.
* Subjects with serum creatinine ≥1.5 mg/dL.
* Is febrile or has other evidence of an infection within 7 days of planned injection.
* Has an allergy or hypersensitivity to chili peppers, capsaicin, or radiographic contrast agents.
* Female subjects who are pregnant, are planning on becoming pregnant, or are currently breastfeeding.
* Subjects with any medical condition that could adversely impact study participation or assessments.
* Subjects who have received new anti-cancer treatments and there is less than one week or four half-lives of the investigational drug, whichever is greater, between the last dose of the new drug and the planned day of IP administration; or had a change in the dose or schedule of the anti-cancer treatments within one week or four half-lives, whichever is greater, between the last dose of the anti-cancer treatment and the planned day of IP administration; or are scheduled to receive a new anti-cancer therapy or investigational product prior to completion of the Day 15 visit.
* Subjects with additional loci of pain above the mid-thoracic level or other pain disorder due to non-cancer etiology, unless both the investigator and the subject are clearly able to distinguish the additional pain from the target pain due to cancer.
* Liver cirrhosis or severe hepatic impairment, with liver function test 3 times above ULN.
* Sensory/peripheral neuropathy of CTCAE Grade 2 or higher.
* Nonstudy related minor surgical procedure ≤5 days or major surgical procedure ≤21 days prior to Screening visit.
* Subjects who have not completely recovered from any toxicities from previous chemotherapy, hormone therapy, immunotherapy, or radiotherapies that are CTCAE Grade 3 or higher.
* Arterial thrombi (including stroke), myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within 3 months prior to Screening visit.
* Corrected QT using Fridericia's formula (QTcF) prolongation.
* Evidence or history of bleeding disorder within 4 weeks prior to IP administration.
* Known HIV or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 3-month
  Grade 3 or 4 Toxicity associated with RTX administration
Maximum tolerated dose (MTD) | 3-month
  Maximum dose without a Grade 3 or 4 toxicity

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Day-28 to Day90 daily
  Daily average pain and daily worst pain on a 0-10 scale

OTHER OUTCOMES:
Daily analgesic consumption (DAC) log | Day-28 to Day90 daily
  Consumption of analgesics compared to baseline
Brief Pain Inventory-Short Form (BPI-SF) | Day-28, Day1, Day2/3, Day8, Day15, Day30, Day60 and Day90
  Quality of life compared to baseline by the total score
Patient Global Impression of Change (PGIC) | Day2/3, Day8, Day15, Day30, Day60 and Day90
  Patient-reported rating of improvement on a 7-point scale, ranking the improvement from (1) to (7), with (1) being no change or worse to (7) being a great deal better and a considerable improvement that has made all the difference.
Modified Numeric Pain Rating Scale (modified NPRS) | Day1, Day2/3, Day8, Day15, Day30, Day60 and Day90
  A 11-point scale for rating average and worst pain at the location intended to be treated with RTX within 12 hours of the clinical visit, with 0 being no pain to 10 being worst pain imaginable.
Modified Brief Pain Inventory-Short Form (modified BPI-SF) | Day1, Day2/3, Day8, Day15, Day30, Day60 and Day90
  Quality of life affected by pain at the location intended to be treated with RTX, each question rates pain level and pain interference on a 0 to 10 scale. For pain level questions, 0 represents no pain and 10 represents pain as bad as can be imagined. For pain interference questions, 0 is "does not interfere" and 10 is "completely interferes".

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (4):
- United States (4):
  - University of Miami/Sylvester Comprehensive Cancer Center, Miami, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Hermann Drive Surgical Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No